CLINICAL TRIAL: NCT06836570
Title: Evalution of the Effects of Platelet Rich Plasma and Low Level Laser Therapy on Postoperative Complications and Wound Healing After Impacted Third Molar
Brief Title: Evalution of the Effects of PRP and LLLT on Postoperative Complications and Wound Healing After Impacted Third Molar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Serap Keskin Tunc, Associate Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YYU-03/18.05.2022
Record Dates: First submitted 2025-01-22; First posted 2025-02-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-01

CONDITIONS: Impacted Third Molar Tooth
Keywords: Platalet rich plasma; Low level laser; impacted third molar
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platalet Rich Plasma (PRP) (Active Comparator): Platelet-rich plasma (PRP) is a preparation of autologous human platelet concentration enriched in a small amount of plasma produced by centrifuging a patient's own blood. It is applied to the extraction socket after the extraction of an impacted wisdom tooth
  Interventions: Biological: Platalet Rich Plasma
- Low Level Laser Therapy (LLLT) (Active Comparator): Low-level laser therapy is a technology that has been used since the mid-1960s to treat a variety of conditions requiring healing stimulation, pain and inflammation relief, and restoration of function. A single 940 nm diode laser was applied intraorally for 120 seconds (BIOLASE) immediately after the extraction and suturing of an impacted wisdom tooth.
  Interventions: Other: Low Level Laser Therapy

INTERVENTIONS:
Biological: Platalet Rich Plasma — Platelet-rich plasma (PRP) is a preparation of autologous human platelet concentration enriched in a small amount of plasma produced by centrifuging a patient's own blood. It is applied to the extraction socket after the extraction of an impacted wisdom tooth.
  Arms: Platalet Rich Plasma (PRP)
Other: Low Level Laser Therapy — Low-level laser therapy is a technology that has been used since the mid-1960s to treat a variety of conditions requiring healing stimulation, pain and inflammation relief, and restoration of function. A single 940 nm diode laser was applied intraorally for 120 seconds (BIOLASE) immediately after the extraction and suturing of an impacted wisdom tooth.
  Arms: Low Level Laser Therapy (LLLT)

SUMMARY:
The aim of the study was to compare the possible effects of platelet-rich plasma (PRP) and low-level laser (BIOLASE) on postoperative complications after extraction of impacted mandibular wisdom teeth. 60 impacted wisdom teeth of 30 healthy individuals who applied to the Department of Oral and Maxillofacial Surgery, Faculty of Dentistry, XXX University, with the indication of extraction of impacted mandibular wisdom teeth were included in the study. 60 impacted wisdom teeth of the individuals were randomly divided into two groups (A and B). In a randomized controlled trial, platelet-rich plasma (PRP) was applied to the first group (A) (one side of the same patients) and low-level laser therapy (LLLT) was applied to the second group (B) (the other side of the same patient) immediately after surgery. VAS (Visual analog scale) for pain assessment, facial measurements for edema assessment and maximum mouth opening for trismus assessment were compared with preoperative values.

DETAILED DESCRIPTION:
The aim of the study was to compare the possible effects of platelet rich plasma (PRP) and low level laser (BIOLASE) on postoperative complications after extraction of impacted lower wisdom teeth. Sixty impacted wisdom teeth of 30 healthy individuals who applied to XXX University, Faculty of Dentistry, Department of Oral, Dental and Maxillofacial Surgery with an indication for extraction of impacted lower wisdom teeth were included in the study. The 60 impacted wisdom teeth of the individuals were randomly divided into two groups (A and B). In a randomised, controlled study, the first group (A) (one side of the same patients) received platelet-rich plasma (PRP) and the second group (B) (the other side of the same patient): diode laser Low-level laser therapy (LLLT) were applied immediately to the patient after surgery. VAS (Visual analogue scale) was used for pain assessment and assessments were made at 3rd, 6th, 12th and 24th hours and at 2nd, 3rd, 4th, 5th, 6th and 7th days. For edema assessment, preoperative facial measurements were repeated on the 2nd and 7th postoperative days and recorded. For trismus evaluation, the maximum mouth opening measurement made preoperatively was repeated and recorded on postoperative days 2 and 7.

ELIGIBILITY:
Inclusion criteria;

* Individuals aged 18 and over,
* Patients with partially impacted wisdom teeth,
* Individuals with systemic status ASA0 and ASA1 according to ASA classification,
* Individuals who have not used any medication in the last two weeks,
* Individuals who do not have a lower second molar missing.

Exclusion criteria;

* Individuals with mouth opening less than 25 mm for various reasons,
* Pregnant and breastfeeding individuals,
* Individuals who do not come to postoperative check-ups,
* Individuals who use different medications other than the recommended medication.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2024-04-23 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 3, 6, 12 and 24 hours and the 2nd, 3rd, 4th, 5th, 6th and 7th days
  In the pain assessment, the patients were given a VAS form at 3, 6, 12 and 24 hours and on the 2nd, 3rd, 4th, 5th, 6th and 7th days and the pain felt by the patient was marked on this scale. This form consists of numbers between 0 and 10. 0 represents 'no pain at all' and 10 represents 'worst possible pain'.
Trismus | preop, 2th and 7th days
  In all patients participating in the study, the maximum interincisal distance for trismus was measured and recorded by the same physician before the operation and on the 2nd and 7th days after the operation.
Edema | preop, 2th and 7th days
  For edema, some anatomical points on the face were taken as reference points and the distance between these points was measured with a tape measure and recorded. The angulus point was determined as the center point and the distances between angulus-tragus, angulus-lateral corner of the eye, angulus-nasal base, angulus-labial commissure and angulus-pogonion point were measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl Üniversitesi Diş Hekimliği Fakültesi, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-01): https://cdn.clinicaltrials.gov/large-docs/70/NCT06836570/Prot_SAP_000.pdf